CLINICAL TRIAL: NCT07247318
Title: The Physiological Effects of Different Non-invasive Respiratory Support in Patients With Acute Hypoxemic Respiratory
Brief Title: The Effects of Different Non-invasive Respiratory Support
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Principal Investigator, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Non-invasive support
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Acute Respiratory Failure (ARF)
MeSH Terms: interventions — Continuous Positive Airway Pressure; Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPAP group (Experimental): Patients will receive continuous positive airway pressure
  Interventions: Device: Continuous Positive Airway Pressure
- NIV group (Experimental): Patients will receive non-invasive ventilation
  Interventions: Device: Non-invasive ventilation
- HFNO group (Experimental): Patients will receive HFNO
  Interventions: Device: High-flow nasal oxygen

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Patients were placed at a 45-degree supine position, and noninvasive ventilation was delivered to the patient through a face mask connected to an ICU ventilator. 2.PEEP was started at 5 cm H2O with a FiO2 of 0.5 at initiation. PEEP and FiO2 were titrated to maintain SpO2 between 94 and 98%, remaining constant for at least 5 min. 3.CPAP was initiated with a first session of at least 4 h, the minimally required duration of noninvasive ventilation was 16 hours per day for at least 2 calendar days. Between noninvasive-ventilation sessions, patients received HFNO.
  Arms: CPAP group
Device: Non-invasive ventilation — Patients were placed at a 45-degree supine position, and noninvasive ventilation was also delivered to the patient through a face mask connected to an ICU ventilator. The mask most appropriate for the patient will be selected and adjusted to minimize leakage and pressure points. 2. The inspiratory positive airway pressure (pressure support plus PEEP) was initiated between 12 and 14 cm H2O, PEEP was started at 5 cm H2O with a FiO2 of 0.5 at initiation. FiO2 was titrated to maintain SpO2 between 94 and 98%, remaining constant for at least 5 min. 3. NIV was initiated with a first session of at least 4 h, the minimally required duration of noninvasive ventilation was 16 hours per day for at least 2 calendar days. Between noninvasive-ventilation sessions, patients received HFNO.
  Arms: NIV group
Device: High-flow nasal oxygen — Oxygen was passed through a heated humidifier (MR850, Fisher and Paykel Healthcare) and applied continuously through large-bore binasal prongs, with a gas flow rate of 50 liters per minute and an FiO2 of 0.5 at initiation. HFNO heating temperature was prespecified at 37°C. 2.FiO2 will be titrated to maintain SpO2 between 94 and 98%, remaining constant for at least 5 min. 3.HFNO was applied for at least 2 calendar days.
  Arms: HFNO group

SUMMARY:
Patients with acute hypoxemic respiratory failure (AHRF) typically present with pathophysiological alterations characterized by the coexistence of respiratory dysfunction and hypoxemia. Respiratory dysfunction leads to dyspnea, increased work of breathing, use of accessory respiratory muscles, and hypercapnia, while gas exchange impairment results in hypoxemia. Studies have shown that hypercapnia, acidosis, and hypoxemia can all enhance inspiratory effort, which further increases negative intrathoracic pressure. In these patients, regional differences in airway resistance and lung compliance are often present, causing redistribution of air within the lungs. This redistribution manifests as gas movement from non-dependent to dependent regions, known as "pendelluft," which amplifies regional alveolar strain and ventilation heterogeneity. This phenomenon becomes more pronounced during noninvasive respiratory support when spontaneous breathing is preserved.

Noninvasive respiratory support strategies mainly include high-flow nasal oxygen (HFNO), noninvasive positive pressure ventilation (NIV), and continuous positive airway pressure (CPAP). HFNO delivers high-flow gas through nasal cannulas, generating a certain level of positive end-expiratory pressure (PEEP) and flushing out anatomical dead space to improve gas exchange, thereby reducing inspiratory effort, lowering the work of breathing, and enhancing oxygenation. NIV, typically using pressure support ventilation (NIV-PSV), is a patient-triggered, pressure-targeted mode that provides inspiratory positive pressure above PEEP. By augmenting tidal volume and reducing inspiratory effort, NIV improves gas exchange; however, leaks may limit the effective delivery of PEEP, and full inspiratory synchronization can increase transpulmonary driving pressure and tidal volume. CPAP, by contrast, delivers a constant positive pressure during both inspiration and expiration. Compared with HFNO, CPAP generates higher PEEP, which facilitates alveolar recruitment and more effectively improves oxygenation. Relative to NIV, CPAP may reduce transpulmonary driving pressure and tidal volume.

Different noninvasive respiratory support strategies exert varying effects on respiratory drive and regional lung strain, leading to differences in the occurrence and magnitude of pendelluft. Physiological studies have suggested that CPAP may offer greater benefits in improving oxygenation and reducing inspiratory effort; however, whether it can mitigate the occurrence and extent of pendelluft remains uncertain. Therefore, this study was conducted to visualize and quantitatively assess pendelluft in real time using electrical impedance tomography (EIT), aiming to verify whether CPAP has a superior effect in reducing pendelluft in patients with AHRF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* PaO₂/FiO₂ ≤ 300 mmHg or SpO₂/FiO₂ ≤ 315 (with SpO₂ ≤ 97%);
* Requiring one of the following respiratory supports:

  1. Noninvasive positive pressure ventilation with PEEP ≥ 5 cmH₂O, or
  2. High-flow nasal oxygen therapy with a flow rate ≥ 30 L/min, or
  3. Conventional oxygen therapy with an oxygen flow ≥ 10 L/min, where FiO₂ is calculated using the formula: FiO₂ = 0.21 + (oxygen flow rate × 0.03).

Exclusion Criteria:

* Received CPAP or NIV for more than 24 hours prior to screening.
* Received invasive mechanical ventilation during the current hospitalization.
* Presence of chronic underlying pulmonary disease, or PaCO₂ ≥ 45 mmHg.
* Presence of cardiogenic pulmonary edema.
* Hemodynamic instability, defined as systolic blood pressure < 90 mmHg or norepinephrine-equivalent dose > 0.3 µg/kg/min.
* Impaired consciousness (GCS ≤ 12).
* Patients requiring urgent intubation, including those with respiratory or cardiac arrest, apnea with loss of consciousness or gasping, or severe hypoxemia (defined as SpO₂ < 90% despite 100% oxygen).
* Contraindications to NIV: cardiac or respiratory arrest, coma, untreated pneumothorax, uncontrollable vomiting, upper airway obstruction, hematemesis or severe facial trauma, or thoracic/abdominal surgery within the past 7 days.
* Contraindications to EIT: implanted cardiac pacemaker, unstable spinal injury or fracture, or open chest trauma.
* Refusal of endotracheal intubation.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Magnitude of Pendelluft | during the first 48 hours
  magnitude of Pendelluft using a software based on electrical impedance tomography monitoring

SECONDARY OUTCOMES:
pH | during the first 48 hours
  Arterial blood gas analysis
Partial pressure of oxygen (PaO2) | during the first 48 hours
  Arterial blood gas analysis
Partial Pressure of Carbon Dioxide (PaCO2) | during the first 48 hours
  Arterial blood gas analysis
Pao2/FiO2 | during the first 48 hours
  Arterial blood gas analysis
Occlusion pressure at 100 ms (P0.1) | during the first 48 hours
  Monitoring with non-invasive ventilator
Occluded inspiratory airway pressure (Pocc) | during the first 48 hours
  Monitoring with a non-invasive ventilator
center of ventilation | during the first 48 hours
  monitoring with EIT
RVD | during the first 48 hours
  Monitoring with EIT

IPD SHARING:
Plan to Share IPD: No